CLINICAL TRIAL: NCT01240980
Title: A Randomized, Double-Blinded, Placebo-Controlled, Ascending Single-Dose Study to Evaluate the Safety, Pharmacokinetics, and Pharmacodynamics of BMS-903452 in Healthy Subjects and Subjects With Type 2 Diabetes Mellitus
Brief Title: Safety Study of BMS-903452 in Healthy Subjects (Panel 1-7) & Relative Bioavailability of the Crystalline and Amorphous Forms of BMS-903452 [Panels 4, 6, 11 & 12(Part A)], and Subjects With Type 2 Diabetes Mellitus (Part B)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MB125-001
Record Dates: First submitted 2010-11-11; First posted 2010-11-15 (Estimated); Last update posted 2012-03-15 (Estimated); Status verified 2011-11

CONDITIONS: Diabetes
MeSH Terms: conditions — Diabetes Mellitus | interventions — 5-chloro-4-((1-(5-chloropyrimidin-2-yl)piperidin-4-yl)oxy)-1-(2-fluoro-4-(methylsulfonyl)phenyl)pyridin-2(1H)-one

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (12):
- BMS-903452 (0.1 mg) or Placebo - A1 (Experimental): (Healthy Subjects)
  Interventions: Drug: BMS-903452; Drug: Placebo
- BMS-903452 (0.6 mg) or Placebo - A2 (Experimental): (Healthy Subjects)
  Interventions: Drug: BMS-903452; Drug: Placebo
- BMS-903452 (3.0 mg) or Placebo - A3 (Experimental): (Healthy Subjects)
  Interventions: Drug: BMS-903452; Drug: Placebo
- BMS-903452 (10 mg) or Placebo - A4 (Experimental): (Healthy Subjects)
  Interventions: Drug: BMS-903452; Drug: Placebo
- BMS-903452 (30 mg) or Placebo - A5 (Experimental): (Healthy Subjects)
  Interventions: Drug: BMS-903452; Drug: Placebo
- BMS-903452 (60 mg) or Placebo - A6 (Experimental): (Healthy Subjects)
  Interventions: Drug: BMS-903452; Drug: Placebo
- BMS-903452 (120 mg) or Placebo - A7 (Experimental): (Healthy Subjects)
  Interventions: Drug: BMS-903452; Drug: Placebo
- BMS-903452 (0.6 mg) or Placebo - B1 (Experimental): (Subjects with type 2 Diabetes Mellitus)
  Interventions: Drug: Placebo; Drug: BMS-903452
- BMS-903452 (10 mg) or Placebo - B2 (Experimental): (Subjects with type 2 Diabetes Mellitus)
  Interventions: Drug: Placebo; Drug: BMS-903452
- BMS-903452 (120 mg) or Placebo - B3 (Experimental): (Subjects with type 2 Diabetes Mellitus)
  Interventions: Drug: Placebo; Drug: BMS-903452
- BMS-903452 (10 mg) or Placebo - A11 (Experimental): (Healthy Subjects)
  Interventions: Drug: BMS-903452; Drug: Placebo
- BMS-903452 (60 mg) or Placebo - A12 (Experimental): (Healthy Subjects)
  Interventions: Drug: BMS-903452; Drug: Placebo

INTERVENTIONS:
Drug: BMS-903452 — Solution, Oral, 0.1 mg, once daily, 1 day
  Arms: BMS-903452 (0.1 mg) or Placebo - A1
Drug: BMS-903452 — Solution, Oral, 0.6 mg, once daily, 1 day
  Arms: BMS-903452 (0.6 mg) or Placebo - A2
Drug: BMS-903452 — Suspension, Oral, 3.0 mg, once daily, 1 day
  Arms: BMS-903452 (3.0 mg) or Placebo - A3
Drug: BMS-903452 — Suspension, Oral, 10 mg, once daily, 1 day
  Arms: BMS-903452 (10 mg) or Placebo - A4
Drug: BMS-903452 — Suspension, Oral, 30 mg, once daily, 1 day
  Arms: BMS-903452 (30 mg) or Placebo - A5
Drug: BMS-903452 — Suspension, Oral, 60 mg, once daily, 1 day
  Arms: BMS-903452 (60 mg) or Placebo - A6
Drug: BMS-903452 — Suspension, Oral, 120 mg, once daily, 1 day
  Arms: BMS-903452 (120 mg) or Placebo - A7
Drug: Placebo — Solution, Oral, 0 mg, once daily, 1 day
  Arms: BMS-903452 (0.1 mg) or Placebo - A1; BMS-903452 (0.6 mg) or Placebo - A2; BMS-903452 (0.6 mg) or Placebo - B1
Drug: Placebo — Suspension, Oral, 0 mg, once daily, 1 day
  Arms: BMS-903452 (10 mg) or Placebo - A4; BMS-903452 (10 mg) or Placebo - B2; BMS-903452 (120 mg) or Placebo - A7; BMS-903452 (120 mg) or Placebo - B3; BMS-903452 (3.0 mg) or Placebo - A3; BMS-903452 (30 mg) or Placebo - A5; BMS-903452 (60 mg) or Placebo - A6
Drug: BMS-903452 — Suspension using crystalline form, Oral, 10 mg, once daily, 1 day
  Arms: BMS-903452 (10 mg) or Placebo - A11
Drug: BMS-903452 — Suspension using crystalline form, Oral, 60 mg, once daily, 1 day
  Arms: BMS-903452 (60 mg) or Placebo - A12
Drug: Placebo — Suspension using crystalline form, Oral, 0 mg, once daily, 1 day
  Arms: BMS-903452 (10 mg) or Placebo - A11; BMS-903452 (60 mg) or Placebo - A12
Drug: BMS-903452 — Solution, Oral, 0.6 mg, once daily, 1 day
  Arms: BMS-903452 (0.6 mg) or Placebo - B1
Drug: BMS-903452 — Suspension, Oral, 10 mg, once daily, 1 day
  Arms: BMS-903452 (10 mg) or Placebo - B2
Drug: BMS-903452 — Suspension, Oral, 120 mg, once daily, 1 day
  Arms: BMS-903452 (120 mg) or Placebo - B3

SUMMARY:
The purpose of this study is to evaluate the safety, tolerability and effect on blood glucose control of BMS-903452 compared to placebo in healthy subjects & relative bioavailability of the crystalline and amorphous forms of BMS-903452 [Panels 4,6,11 & 12(Part A)] ; and subjects with type 2 Diabetes Mellitus (Part B). The study will also determine the amount of BMS-903452 in the blood.

ELIGIBILITY:
Inclusion Criteria:

* Clinically healthy or Clinical diagnosis of Type 2 diabetes on a stable dose of metformin monotherapy

Exclusion Criteria:

* Type 1 Diabetes
* History of significant heart disease
* Prior bariatric surgery
* Women of childbearing potential

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 104 (Actual)
Dates: Start 2010-11; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Safety and Tolerability of the investigational drug, as assessed by adverse event monitoring, physical examinations, clinical laboratory determinations, electrocardiograms (ECG), and vital sign assessments | Within 10 days of study drug administration

SECONDARY OUTCOMES:
Pharmacodynamic activity of the investigational drug on glucose and hormones regulating glucose metabolism | Within 2 days of study drug administration
Effect on electrocardiographic (ECG) parameters | Within 10 days of study drug administration
Percent urinary recovery (% UR) | Within 10 days of study drug administration
  derived by non-compartmental methods by a validated pharmacokinetic program. Actual times will be used for the analyses
Renal clearance (CLR) from plasma | Within 10 days of study drug administration
  derived by non-compartmental methods by a validated pharmacokinetic program. Actual times will be used for the analyses
The single-dose pharmacokinetics parameter maximum observed concentration in plasma (Cmax) of BMS-903452 will be derived from the plasma concentration versus time data | Within 10 days after study drug administration
The single-dose pharmacokinetics parameter time to reach maximum observed concentration in plasma (Tmax) of BMS-903452 will be derived from the plasma concentration versus time data | Within 10 days after study drug administration
The single-dose pharmacokinetics parameter time Area under the plasma concentration-time curve from time zero extrapolated to infinity AUC(INF) of BMS-903452 will be derived from the plasma concentration versus time data | Within 10 days after study drug administration
The single-dose pharmacokinetics parameter Area under the plasma concentration-time curve from time zero to last measurable sampling time AUC (0-T) of BMS-903452 will be derived from the plasma concentration versus time data | Within 10 days after study drug administration
The single-dose pharmacokinetics parameter Terminal-phase elimination half-life in plasma (T-Half) of BMS-903452 will be derived from the plasma concentration versus time data | Within 10 days after study drug administration
The single-dose pharmacokinetics parameter apparent clearance from plasma after extra-vascular administration (CLT/F) of BMS-903452 will be derived from the plasma concentration versus time data | Within 10 days after study drug administration

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (2):
- United States (2):
  - Comprehensive Phase One, Miramar, Florida
  - Ppd Development, Lp, Austin, Texas

REFERENCES:
- See also: Investigator Inquiry form — http://www.bms.com/clinical_trials/Pages/Investigator_Inquiry_form.aspx